CLINICAL TRIAL: NCT06631820
Title: The Effect of the Nutraceutical (-)- Epicatechin on Myosteatosis in Patients With Advanced CKD: a Pilot Study (EPIC-CKD)
Brief Title: The Effect of the Nutraceutical (-)- Epicatechin on Myosteatosis in Patients With Advanced CKD
Acronym: EPIC-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Alice Sabatino, Research Specialist, Karolinska Institutet
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-04198-01
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease(CKD); Myosteatosis; Mitochondrial Dysfunction; Muscle Function; Muscle Mass
Keywords: myosteatosis; epicatechin; nutraceuticals; chronic kidney disease; mitochondrial dysfunction; muscle regeneration; muscle function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Mitochondrial Diseases | interventions — Catechin

STUDY DESIGN:
Intervention Model Description: This is a pilot treatment crossover interventional trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control phase (No Intervention): patients will undergo 8 weeks without the supplement after enrolment to allow for a control phase
- experimental phase (Experimental): after 8 weeks of control phase, patients will receive the supplement for 8 weeks
  Interventions: Dietary Supplement: Epicatechin extract

INTERVENTIONS:
Dietary Supplement: Epicatechin extract — In the experimental phase, patients will take 50 mg of (-)- Epicatechin twice a day for 8 weeks (total dose 100mg/day). The nutraceutical will be supplied as monodose sachets from Aayam Therapeutics.Study participants will mix the sachet powder with juice (10-20mL) in the morning 15 minutes before breakfast and in the evening 15 minutes before sleeping or 1h after dinner.
  Arms: experimental phase

SUMMARY:
Some foods have components that can prevent and treat some diseases and provide beneficial effects for health. These components naturally occurring in foods are called nutraceuticals. Recently, it was found that Epicatechin, which is a kind of nutraceutical from the Catechin's family naturally occurring in green tea and cocoa, has positive effects on muscle mass and strength of people with chronic diseases.

People with chronic kidney disease often present muscle loss and lack of strength that are not easily treated with regular diet and physical activity. We here propose a study where 10 individuals with chronic kidney disease will receive a dose of Epicatechin for 8 weeks and we aim to test if Epicatechin improves general muscle health. Based on what is known, we expect to see an increase in muscle mass and strength.

The dose of Epicatechin provided (100 mg/day) is safe, since it is much lower than the dose usually available in supplements. In addition, this is the form naturally present in green tea and cocoa and in similar amounts. Subjects participating in the study will be evaluated for muscle mass and strength three times during the study. Muscle mass and muscle quality will be evaluated by ultrasound and magnetic resonance imaging. The participants will also perform some tests like walking in a corridor and seating and standing from a chair to measure their strength and performance. Adverse side effects will be monitored via telephone, and safety will be assessed by monthly blood tests that will evaluate liver and kidney function. If this study shows that Epicatechin can promote muscle growth and strength, it will positively affect patients with chronic kidney disease that might benefit of a natural substance from food to improve muscle health.

DETAILED DESCRIPTION:
The effect of ageing and chronic diseases on the skeletal muscle is of great interest for studies in clinical nutrition. In the setting of chronic kidney disease (CKD), CKD-related metabolic alterations act synergistically with other risk factors in the deterioration of muscle health. Loss of muscle mass and the replacement of contractile muscle fibers by adipose tissue (i.e. myosteatosis) have been shown to decrease muscle strength and function and have a negative effect on patient centred outcomes, such as quality of life.

Considering that patients with low strength have an increased risk of falling, less independency to perform routine tasks and are more vulnerable to stressors with increased risk for recurring hospitalizations, infections, and mortality, it is of utmost importance to explore treatment strategies to overcome muscle abnormalities while improving function. Recently, interventional trials using the nutraceutical (-)- Epicatechin, an abundant flavanol present in cacao and green tea, showed an increase in skeletal muscle mass and exercise capacity through stimulating mitochondrial biogenesis. On this regard, this pilot study aims to evaluate if 100mg of (-)- Epicatechin can help ameliorate muscle abnormalities in patients with CKD.

Aims: This study aims:

1. To evaluate the effect of nutraceutical (-)- Epicatechin on myosteatosis and functional capacity of patients with advanced CKD.
2. To evaluate the effect of nutraceutical (-)- Epicatechin on markers of muscle regeneration.
3. To evaluate the effect of nutraceutical (-)- Epicatechin on markers of mitochondrial dysfunction

This project is a feasibility pilot study to test the effect of the nutraceutical (-)- Epicatechin on muscle health. To allow for a control phase, this study has a cross-over with open label design. We here describe the methodological approach that will allow us to achieve the proposed aims.

Patients will be pre-selected from medical records and contacted telephonically by the investigators to be invited to participate, if they accept, they will be invited to come to the research center to receive an explanation regarding the study, sign the informed consent and undergo a screening visit.

Sample size estimation: In this pilot study, we will utilize a convenience sample of 10 subjects.

Study design and intervention After enrolment, patients will be followed for 8 weeks without receiving the nutraceutical. After this control period, patients will take 50 mg of (-)- Epicatechin twice a day for 8 weeks (total dose 100mg/day). The nutraceutical will be supplied as monodose sachets from Aayam Therapeutics.Study participants will mix the sachet powder with juice (10-20mL) in the morning 15 minutes before breakfast and in the evening 15 minutes before sleeping or 1h after dinner.

The study will comprise 5 visits in total. The first visit will be a screening visit. During the screening visit patients will be oriented to not change their diets during the study period and they will be instructed on how to collect 24h urine to bring at the baseline visit. After 1-2 weeks patients will come back for the baseline visit (visit 1) when they will undergo all evaluations and sampling as described below.The interval between first and second visit is of 8 weeks. At week 8 (visit 2), patients will undergo all study evaluations and sampling, will bring another 24h urine collection and will receive the supplements to be used in the next 8 weeks. After 4 weeks receiving the supplement, patients will receive a phone call (visit 3) to enquire about gastrointestinal symptoms and to be invited to go to their local vårdcentral to perform the safety blood tests (see below). After another 4 weeks patients will come back for the end-of -study visit (visit 4), in which they will perform all study evaluations and sampling again.

The evaluation at patient's local vårdcentral can take place any day during the selected week, while the end-of-study visit must take place within 1 week of the end of week 16 (see detailed picture below).

The duration of the 3 main visits is expected to be 3-4h, patients will receive food after blood collection in a fasting state.

Study variables:

Clinical and demographic variables: age, sex, Charlson comorbidity index, aetiology of the nephropathy will be recorded at baseline visit.

Nutritional and body composition assessment: nutritional evaluation will be performed at baseline, week 8 and week 16.

* Anthropometric variables: Body weight, height, waist circumference, calf circumference.
* Body composition variables:

Total body skeletal muscle and phase angle will be measured with bioimpedance analysis.

Myosteatosis and skeletal muscle quantity of patients will be assessed with 2 imaging modalities: Magnetic Resonance Imaging (MRI) and Ultrasound (US). MRI and US will be used to assess the level of myosteatosis and markers of muscle mass of the quadriceps muscle. US's reliability and validity in assessing muscle quantity and myosteatosis will be studied in comparison to MRI.

Measurements will be performed at the mid-point between the upper pole of the patella and the anterior superior iliac spine in the dominant leg. US will be performed before the MRI and a vitamin D pill will be used to marc the spot for the MRI assessment.

* US: We will use a B-mode wall tracking US device (Clarius, Vancouver, Canada) already available at the research center of Karolinska Institute. Measurements will be performed by a researcher with extensive experience in assessing body composition by using US and will follow a standardized protocol applied repeatedly in patients with acute and chronic kidney disease. Measurements don't take more than 10 minutes. All images will be stored anonymously, and measurements will be performed afterwards by using the software ImageJ (https://imagej.nih.gov/ij/index.html). Two muscles will be identified, the rectus femoris and vastus intermedius. The collected images will allow us to measure muscle thickness, rectus femoris cross-sectional area, rectus femoris and vastus intermedius echogenicity. While thickness and cross-sectional area provide information on muscle quantity, the echogenicity of the muscle provides information on myosteatosis.
* MRI: We will evaluate rectus femoris volume, rectus femoris and vastus intermedius thickness, and rectus femoris cross-sectional area to evaluate muscle quantity. Myosteatosis will be evaluated by applying quantitative fat water imaging (Dixon imaging), information on intermuscular adipose tissue (IMAT), intramuscular adipose tissue, and average myosteatosis level will be performed by experienced radiologist.

Functional tests: Strength will be assessed by handgrip strength using a portable dynamometer, and by the chair stand test (5 time sit to stand and 30 seconds sit-to stand test). Performance will be assessed by the gait speed test, that evaluates the normal speed that a person usually walks and by the 6 minutes walking distance test. An integrated functional test called Short Physical Performance Battery (SPPB), will be used (at baseline, week 8 and week.

Safety assessment: Monitoring will occur at baseline, week 8 (in person visit), week 12 (by phone call and local vårdcentral for exams), and week 16 (in person visit). Safety will be assessed by frequent monitoring of adverse events, gastrointestinal symptoms, and blood parameters (i.e. aspartate aminotransferase [ASAT], alanine aminotransferase [ALAT] and serum creatinine).

Laboratorial data For the screening visit, after signing the informed consent patients will undergo blood sampling for assessment of serum creatinine and liver function.

At study baseline, week 8 and week 16 patients will perform the following blood tests in a 8h fasting state: serum creatinine, ASAT/ALAT, glycemia, HbA1c, total cholesterol, uric acid, PTH, free testosterone, LDL cholesterol, HDL cholesterol, Triglycerides, and CRP.

Blood samples will be stored for posterior evaluation of oxidative stress markers [protein carbonylation, 8-hydroxy-2'-deoxyguanosine [8-OhdG]]), epigenetic clock (DNA metilation clocks evaluation), microbial DNA (as an exploratory analysis to assess the effect of epicatechin on gut microbiota), and specific markers that will allow us to achieve aims 2 and 3 (see below).

Markers to evaluate aim 2: blood markers that signals for muscle regeneration are myostatin, follistatin and GDF-11.

Markers to evaluate aim 3: blood markers that evaluate mitochondrial dysfunction include lactate, pyruvate, mitochondrial copy numbers, creatine phosphokinase, FGF-21, GDF-15.

Patients will also bring a 24h urine sample from the day before the visit to measure urinary urea nitrogen, sodiuria, calciuria and oxaluria. The urine sample will not be stored.

Data on patients' medication will be collected at every main visit, with special attention to erythropoietin usage. Patients will also receive an activity monitor at baseline to be used during the entire study period.

Adherence will be evaluated based on the supplement's leftovers at the end of the study.

Significance:

To treat sarcopenia and myosteatosis in CKD is a challenge. Patients with advanced CKD have anabolic resistance which is defined by a reduced stimulation in muscle protein synthesis after anabolic stimuli, such as exercise and dietary protein, and is also a feature of mitochondrial dysfunction. This project innovates by testing a nutraceutical available in various food sources, but especially in cacao and green tea, that could help overcome this condition of anabolic resistance. If our hypotheses are confirmed, the nutraceutical (-)- Epicatechin could be used as an adjuvant factor in the treatment of sarcopenia and myosteatosis in patients with advanced CKD.

ELIGIBILITY:
Inclusion Criteria:

* estimated glomerular filtration rate (eGFR) < 29 ml/min/1.75m2
* no chronic or acute known liver disease
* not intended to initiate renal replacement therapy treatment in the next 4 months according to nephrologist clinical judgment

Exclusion Criteria:

* signs of active infection
* acute vasculitis
* type 1 diabetes
* use of steroids medication
* transplanted patients
* patients with deambulatory impairment (wheelchair users, bed rest)
* patients on compassionate care for the end of life
* with advanced neurological disorders
* with cognitive impairments
* with active cancer diagnosis
* participation in another interventional trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Epicatechin supplementation effect on myosteatosis | At enrolment, at 8 weeks from enrolment and at 16 weeks from enrolment.
  Myosteatosis will be evaluated by Ultrasound (US) and Magnetic resonance imaging (MRI).
  US: We will use a B-mode wall tracking US device (Clarius, Vancouver, Canada).Two muscles will be identified, the rectus femoris and vastus intermedius. The collected images will allow us to measure muscle thickness, rectus femoris cross-sectional area, rectus femoris and vastus intermedius echogenicity. While thickness and cross-sectional area provide information on muscle quantity, the echogenicity of the muscle provides information on myosteatosis.
  MRI: We will evaluate rectus femoris volume, rectus femoris and vastus intermedius thickness, and rectus femoris cross-sectional area to evaluate muscle quantity. Myosteatosis will be evaluated by applying quantitative fat water imaging (Dixon imaging), information on intermuscular adipose tissue (IMAT), intramuscular adipose tissue, and average myosteatosis level will be performed by experienced radiologist.
Epicatechin supplementation effect on muscle function | At enrolment, at 8 weeks from enrolment and at 16 weeks from enrolment.
  Functional tests: Strength will be assessed by handgrip strength using a portable dynamometer, and by the chair stand test (5 time sit to stand and 30 seconds sit-to stand test). Performance will be assessed by the gait speed test, that evaluates the normal speed that a person usually walks and by the 6 minutes walking distance test. An integrated functional test called Short Physical Performance Battery (SPPB), will be used (at baseline, week 8 and week 16).

SECONDARY OUTCOMES:
Epicatechin supplementation effect on markers of muscle regeneration | At enrolment, at 8 weeks from enrolment and at 16 weeks from enrolment.
  We will evaluate the following blood markers that are indicators of muscle regeneration: myostatin, follistatin and GDF-11.
Epicatechin supplementation effect on markers of mitochondrial dysfunction | At enrolment, at 8 weeks from enrolment and at 16 weeks from enrolment.
  Mitochondrial dysfunction will be evaluated by applying the following blood markers: lactate, pyruvate, mitochondrial copy numbers, creatine phosphokinase, FGF-21, GDF-15.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

REFERENCES:
- [Background] Gamboa JL, Roshanravan B, Towse T, Keller CA, Falck AM, Yu C, Frontera WR, Brown NJ, Ikizler TA. Skeletal Muscle Mitochondrial Dysfunction Is Present in Patients with CKD before Initiation of Maintenance Hemodialysis. Clin J Am Soc Nephrol. 2020 Jul 1;15(7):926-936. doi: 10.2215/CJN.10320819. Epub 2020 Jun 26. PMID 32591419
- [Background] Gamboa JL, Billings FT 4th, Bojanowski MT, Gilliam LA, Yu C, Roshanravan B, Roberts LJ 2nd, Himmelfarb J, Ikizler TA, Brown NJ. Mitochondrial dysfunction and oxidative stress in patients with chronic kidney disease. Physiol Rep. 2016 May;4(9):e12780. doi: 10.14814/phy2.12780. PMID 27162261
- [Background] Avesani CM, de Abreu AM, Ribeiro HS, Brismar TB, Stenvinkel P, Sabatino A, Lindholm B. Muscle fat infiltration in chronic kidney disease: a marker related to muscle quality, muscle strength and sarcopenia. J Nephrol. 2023 Apr;36(3):895-910. doi: 10.1007/s40620-022-01553-0. Epub 2023 Jan 31. PMID 36719556
- [Background] McDonald CM, Ramirez-Sanchez I, Oskarsson B, Joyce N, Aguilar C, Nicorici A, Dayan J, Goude E, Abresch RT, Villarreal F, Ceballos G, Perkins G, Dugar S, Schreiner G, Henricson EK. (-)-Epicatechin induces mitochondrial biogenesis and markers of muscle regeneration in adults with Becker muscular dystrophy. Muscle Nerve. 2021 Feb;63(2):239-249. doi: 10.1002/mus.27108. Epub 2020 Dec 16. PMID 33125736
- [Background] Taub PR, Ramirez-Sanchez I, Ciaraldi TP, Gonzalez-Basurto S, Coral-Vazquez R, Perkins G, Hogan M, Maisel AS, Henry RR, Ceballos G, Villarreal F. Perturbations in skeletal muscle sarcomere structure in patients with heart failure and type 2 diabetes: restorative effects of (-)-epicatechin-rich cocoa. Clin Sci (Lond). 2013 Oct;125(8):383-9. doi: 10.1042/CS20130023. PMID 23642227